CLINICAL TRIAL: NCT05275231
Title: Better Together: A Patient-centered Approach to Improve Diabetes Among Immigrant Communities
Brief Title: Better Together Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Megha Kumudchandra Shah, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000967; 1K23MD015088-01 (NIH)
Record Dates: First submitted 2022-01-31; First posted 2022-03-11 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes
Keywords: Immigrant; South Asian born Immigrant; African born Immigrant; Social Contact
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dyads (Experimental): This is a pragmatic, pre-post, pilot study. Participants will meet in groups of 12 for the SMA intervention at the conference room at the Emory Family Medicine Center in Dunwoody, Georgia. The intervention will consist of bi-weekly sessions over a 16-week period, with phone check-ins for the remaining weeks. Each session will last 60-90 minutes, and participants will engage in a total of 6 televisit sessions. Sessions will consist of a group-based program for all participants, followed by a personalized care plan, led by a physician. In this dyad-based group, participant's social partner must commit to attend all in-person sessions.
  Interventions: Behavioral: Intensive lifestyle interventions (ILIs)
- Men Only (Active Comparator): This is a pragmatic, pre-post, pilot study. Participants will meet in groups of 12 for the SMA intervention at the conference room at the Emory Family Medicine Center in Dunwoody, Georgia. the intervention will consist of bi-weekly sessions over a 16-week period, with phone check-ins for the remaining weeks. Each session will last 60-90 minutes, and participants will engage in a total of 6 televisit sessions. Sessions will consist of a group-based program for all participants, followed by a personalized care plan, led by a physician. In this group just the participant will receive the intervention.
  Interventions: Behavioral: Intensive lifestyle interventions (ILIs)

INTERVENTIONS:
Behavioral: Intensive lifestyle interventions (ILIs) — Intensive lifestyle interventions (ILIs) is a group-based programs designed to promote weight loss through a combination of diet, activity, and behavior change, decrease Type 2 Diabetes (T2D) incidence in people with prediabetes and reduced complications among people with T2D.

SUMMARY:
This study (Aim 1) seeks to test that a culturally-tailored lifestyle intervention is feasible and acceptable for immigrant men from South Asia and West Africa. This will be a pre-post pilot study of a 16-week lifestyle program for South Asians and West Africans with prediabetes or diabetes in Atlanta. Patients will participate in health-professional-led group visits every other week focused on improving dietary and exercise practices to reduce weight. Groups will be followed at baseline, 4 months and 12 months. Groups will be separated by region of origin (i.e. separate groups for South Asians and West Africans). For Aim 2,the study team will assess intervention spillover effects among participant's self-identified social networks. The study team will ask participants in Aim 1 to name 5 people in their social networks to participate in a survey of health behaviors at baseline and 12-months to assess health behavior practices.

DETAILED DESCRIPTION:
South Asians and Africans are growing immigrant groups at high risk for diabetes in the US. South Asian (SA) (ancestry originating from India, Pakistan, Bangladesh and other parts of South Asia) and Sub-Saharan African immigrant groups make up two of the fastest growing immigrant groups in the US. SAs have higher rates of T2D and cardiovascular disease than whites. Furthermore, SAs without diabetes have a high prevalence of T2D risk factors.

Sub-Saharan African-born immigrants (the proposed study will focus on West African (WA) countries: those originating from Benin, Burkina Faso, Cape Verde, The Gambia, Ghana, Guinea, Guinea-Bissau, Ivory Coast, Liberia, Mali, Mauritania, Niger, Nigeria, Senegal, Sierra Leone, and Togo), whose population in the US has doubled every decade since 1980, are also at high risk for T2D. Dietary patterns of African immigrants are high in carbohydrates and animal protein, compared to African populations who did not immigrate.

These findings in SA and African immigrant communities challenge the well-accepted "healthy immigrant effect" phenomenon (that immigrants are on average healthier than native-born persons), suggesting that more tailored T2D prevention and management strategies are greatly needed to narrow the disparities in outcomes between these and other US populations. Previous trials showed that intensive lifestyle interventions (ILIs), group-based programs designed to promote weight loss through a combination of diet, activity, and behavior change, decrease T2D incidence in people with prediabetes and reduced complications among people with T2D. Additional analyses have shown that the effects of lifestyle interventions are long-lasting, even when participants gain back some of the weight lost during the program.

Family and social networks could be an important factor to improve patient activation, especially for South Asian and African immigrant men. Social networks, defined as someone with social or family ties to an individual, affect health through myriad mechanisms including social support, social influence, social engagement, and access to resources. This study aims to focus on SA and WA immigrant men as model populations to examine preferences, feasibility, and acceptability for a shared medical appointment (SMA) intervention based in primary care and developed with user-driven input and changes in healthy lifestyle practices among participants' social networks. This will be a pre-post pilot study of a 16-week lifestyle program for the mentioned immigrant groups with prediabetes or diabetes in Atlanta. Patients will participate in health-professional-led group visits every other week focused on improving dietary and exercise practices to reduce weight. Groups will be followed at baseline, 4 months and 12 months. For Aim 2, the study team will assess intervention spillover effects among participant's self-identified social networks. The study team will ask participants in Aim 1 to name 5 people in their social networks to participate in a survey of health behaviors at baseline and 12-months to assess health behavior practices.

ELIGIBILITY:
Inclusion Criteria for Aim 1:

* Men >18 years of age
* Diagnosis of Type 2 Diabetes (T2D) (documented A1c of ≥ 5.7% or fasting blood glucose of >100) or prediabetes
* A family member or peer is willing to participate and attend all sessions as a social partner (if enrolling in dyad arm)
* Proficiency in English(if in dyad, at least one member of each dyad)
* Willingness to provide written consent

Inclusion Criteria for Aim 2:

* Proficient in English
* Age greater than or equal to 18 years

Exclusion Criteria Aim 1 and 2:

* Type 1 diabetes or diabetes secondary to other conditions (e.g. steroid-induced, pancreatic insufficiency, or chemotherapy-induced)
* Malignancy or life-threatening illness with life expectancy of <5 years
* End-stage disease or serious illness that prohibits participation (e.g. end-stage renal disease or class IV congestive heart failure)
* Inability to perform unsupervised physical activity
* Diagnosed with cognitive deficits or limited decision-making capacity
* Alcohol or substance abuse
* Homelessness or no fixed address.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megha Shah, MD, Principal Investigator — Emory University
Locations (1):
- Emory Family Medicine Center, Dunwoody, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Any de-identified data, upon request
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available 6 months after data collection is complete
Access Criteria: De-identified Data will be available to any party who completes a data use agreement that describes for what purpose the data will be used with a clear analysis plan.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Emory Family Medicine Center. Participant enrollment began on April 4, 2022, and all follow-up assessments were completed by January 1, 2024 The study was a quasi-experimental design to understand preferences in this community. The PI offered a men-only group with very little interest in this group thus this arm was never carried forward. No subjects were enrolled in this group. Men-only group was not supposed to be a comparator arm.
Period: Overall Study
Arm/Group | Dyads
Started | 54 (54 dyads or 108 total)
Completed | 54
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: No baseline characteristics data was collected on the support group.
Groups:
- Participants: Participants who co-participated in a 5-session lifestyle intervention for diabetes management and prevention
- Support Group: Support group comprised of participant's social partner.
- Total: Total of all reporting groups
Arm/Group | Participants | Support Group | Total
Number analyzed (Participants) | 54 | 54 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: No baseline characteristics were collected from support group
  years
    number analyzed (Participants) | 54 | 0 | 54
    (all) | 52.8 (10.5) |  | 52.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants] — The initial plan was to recruit Males only, but due to recruiting challenges faced during COVID, the PI included Women in the study as well. Population: No baseline characteristics were collected on this group
  Participants
    number analyzed (Participants) | 54 | 0 | 54
    Female | 28 |  | 28
    Male | 26 |  | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Native Language [Count of Participants; unit: Participants] — Population: No baseline characteristics were collected on this group
  Participants
    Bengali: number analyzed (Participants) | 54 | 0 | 54
    Bengali | 53 |  | 53
    Other: number analyzed (Participants) | 54 | 0 | 54
    Other | 1 |  | 1
English Fluency [Count of Participants; unit: Participants] — Population: No baseline characteristics were collected on this group
  Participants
    Very good: number analyzed (Participants) | 54 | 0 | 54
    Very good | 13 |  | 13
    Good: number analyzed (Participants) | 54 | 0 | 54
    Good | 21 |  | 21
    Not good: number analyzed (Participants) | 54 | 0 | 54
    Not good | 16 |  | 16
    Not good at all: number analyzed (Participants) | 54 | 0 | 54
    Not good at all | 4 |  | 4
Language Spoken at Home [Count of Participants; unit: Participants] — Population: No baseline characteristics were collected from support group
  Participants
    Mostly English: number analyzed (Participants) | 54 | 0 | 54
    Mostly English | 0 |  | 0
    Mix of English/ Native: number analyzed (Participants) | 54 | 0 | 54
    Mix of English/ Native | 10 |  | 10
    Mostly Native: number analyzed (Participants) | 54 | 0 | 54
    Mostly Native | 43 |  | 43
    Other: number analyzed (Participants) | 54 | 0 | 54
    Other | 1 |  | 1
Education [Count of Participants; unit: Participants] — Population: No baseline characteristics were collected from support group
  Participants
    Some high school: number analyzed (Participants) | 54 | 0 | 54
    Some high school | 8 |  | 8
    High School Graduate: number analyzed (Participants) | 54 | 0 | 54
    High School Graduate | 5 |  | 5
    Some College: number analyzed (Participants) | 54 | 0 | 54
    Some College | 5 |  | 5
    unknown: number analyzed (Participants) | 54 | 0 | 54
    unknown | 36 |  | 36
Employment Status [Count of Participants; unit: Participants] — Population: No baseline characteristics were collected from support group
  Participants
    Employed for wages: number analyzed (Participants) | 54 | 0 | 54
    Employed for wages | 24 |  | 24
    Self-employed: number analyzed (Participants) | 54 | 0 | 54
    Self-employed | 1 |  | 1
    Homemaker: number analyzed (Participants) | 54 | 0 | 54
    Homemaker | 11 |  | 11
    Student: number analyzed (Participants) | 54 | 0 | 54
    Student | 1 |  | 1
    Retired: number analyzed (Participants) | 54 | 0 | 54
    Retired | 13 |  | 13
    Unemployed: number analyzed (Participants) | 54 | 0 | 54
    Unemployed | 4 |  | 4
Marital Status [Count of Participants; unit: Participants] — No baseline characteristics were collected from support group Population: No baseline characteristics were collected from support group
  Participants
    Married: number analyzed (Participants) | 54 | 0 | 54
    Married | 45 |  | 45
    Divorced: number analyzed (Participants) | 54 | 0 | 54
    Divorced | 1 |  | 1
    Widowed: number analyzed (Participants) | 54 | 0 | 54
    Widowed | 7 |  | 7
    unknown: number analyzed (Participants) | 54 | 0 | 54
    unknown | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Group Preference
Description: Which group of the study are participants choosing between the single participant group or the dyad.
  Preferences will be assessed by quantifying number enrolled in each group.
Time Frame: Baseline
Population: No data was collected from the support group for this Outcome measure.
Measure: Number; unit: participants
Arm/Group | Dyads | Men Only
Number analyzed (Participants) | 54 | 0
participants | 54 |

2. Primary Outcome: Feasibility: Proportion of Subjects Who Enroll
Description: The proportion of adults who are contacted and informed about the study and who enroll during study baseline. Feasibility will be assessed by quantifying rate of enrollment, number of sessions attended by participants (for dyad arm, will assess participant and social contact, individually and together).
Time Frame: Baseline
Population: No data was collected on the support group for this outcome measure. 122 is the number of people who were approached for the study.
Measure: Number; unit: participants enrolled
Arm/Group | Dyads
Number analyzed (Participants) | 122
participants enrolled | 54

3. Primary Outcome: Retention: Number of Sessions Attended
Description: Number of sessions attended; for dyads, this would include sessions attended together and separately, over the 16-week study period.
  There were 5 sessions total.
Time Frame: From baseline to week 16
Population: The data collected for this outcome is only for the sessions attended together.
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | Participants
Number analyzed (Participants) | 54
sessions | 4.7 (0.53)

4. Primary Outcome: Acceptability: Satisfaction Questionnaire
Description: Questionnaires assessed participant perceptions of ILI after the program to evaluate satisfaction with the program and suggestions for program improvement.
  Acceptability will be assessed by quantifying Likert-like scales of satisfaction of overall intervention. This is a 0 to 5 scale, where "0" represents the least level of satisfaction and "5" represents the highest level of satisfaction.
Time Frame: Month 6
Population: No data was collected from the support group for this Outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants
Number analyzed (Participants) | 54
score on a scale | 5 (0)

5. Other Pre Specified Outcome: Changes in Body Mass Index (BMI)
Description: Participant's weight will be measured in kilograms using a calibrated, standardized scale, and height will be measured in meters (m), using a standardized stadiometer. BMI will be calculated using the standard formula of kg/m^2.
Time Frame: Baseline, month 6
Population: No data was collected from the support group for this Outcome measure.
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Participants
Number analyzed (Participants) | 53
kg/m2
  Baseline | 26.56 (3.71)
  Month 6 | 25.92 (4.94)

6. Other Pre Specified Outcome: Changes in Abdominal Waist Circumference
Description: Waist circumference will be measured in centimeters (cm) by the World Health Organization recommended method.
Time Frame: Baseline, month 6
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Changes in Diastolic Blood Pressure
Description: Participant's systolic and diastolic blood pressure will be measured using standard procedures with a manual cuff.
  Diastolic blood pressure is the amount of pressure in the arteries when the heart is at rest between beats. Current guidelines identify normal diastolic blood pressure as lower than 80 mmHg.
Time Frame: Baseline, month 6
Population: No data was collected from the support group for this Outcome measure.
Measure: Mean (Standard Deviation); unit: mm of HG
Arm/Group | Participants
Number analyzed (Participants) | 52
mm of HG
  Baseline | 76.32 (7.65)
  Month 6 | 76.0 (7.5)

8. Other Pre Specified Outcome: Changes in Hemoglobin A1c
Description: Participant's Hemoglobin A1c (HbA1c) will be measured with a point-of-care testing (POCT) well-validated clinical instrument. Normal values for HbA1c are below 5.7% while values of 6.5% and above indicate diabetes.
Time Frame: Baseline, month 6
Population: No data was collected from the support group for this Outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of HbA1C
Arm/Group | Participants
Number analyzed (Participants) | 51
percentage of HbA1C
  Baseline | 7.57 (1.49)
  Month 6 | 6.72 (0.81)

9. Other Pre Specified Outcome: Changes in Body Weight
Description: Participant's weight will be measured in kilograms using a calibrated, standardized scale.
Time Frame: Baseline, month 6
Population: No data was collected from the support group for this Outcome measure.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Participants
Number analyzed (Participants) | 54
pounds
  Baseline | 155.4 (25.96)
  Month 6 | 152.8 (25.60)

10. Other Pre Specified Outcome: Changes in Systolic Blood Pressure
Description: Participant's systolic and diastolic blood pressure will be measured using standard procedures with a manual cuff.
  Systolic blood pressure is the amount of pressure the heart generates when pumping blood through the arteries to the body. Current guidelines identify normal systolic blood pressure as lower than 120 mmHg.
Time Frame: Baseline, month 6
Population: No data was collected from the support group for this Outcome measure.
Measure: Mean (Standard Deviation); unit: mm of Hg
Arm/Group | Participants
Number analyzed (Participants) | 52
mm of Hg
  Baseline | 129.7 (19.40)
  Month 6 | 123.9 (13.95)

11. Other Pre Specified Outcome: Changes in Physical Activity
Description: Participants will be asked to keep a daily activity log (minutes of exercise performed daily will be logged). All logged exercises will be considered physical activity. The study coordinators will measure the amount in hours of exercise performed and compare each participant's log at the different time points to asses in that subject's physical activity
Time Frame: Baseline, month 6
Population: No data was collected from the support group for this Outcome measure.
Measure: Mean (Standard Deviation); unit: minutes/ week
Arm/Group | Participants
Number analyzed (Participants) | 54
minutes/ week
  Baseline | 130.7 (187.8)
  Month 6 | 245.5 (154.9)

12. Other Pre Specified Outcome: Changes in Diet
Description: Changes in diet will be measured using the Rapid Eating and Activity Assessment for Participants short version (REAP-S).
  The REAP-S consists of 13 scored questions. Responses of 'usually/often' receive 1 point, 'sometimes' receives 2 points, and 'rarely/never or does not apply to me' receives 3 points. Possible scores ranged from 13 to 39 with a higher score indicating a higher diet quality.
Time Frame: Baseline, month 6
Population: The average was collected by analyzing the points scored on each item (points rated 1-3).
  No data was collected from the support group for this Outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants
Number analyzed (Participants) | 54
score on a scale
  Baseline | 2.140 (1.3)
  Month 6 | 2.05 (1.31)

13. Other Pre Specified Outcome: Change in Weight Control Strategies Scale (WCSS) Score for Social Contacts
Description: Participants' social contacts will complete the WCSS. The WCSS is a 30-item questionnaire asking about weight control practices. Responses are given on a 5-point scale when 0 = never and 4 = always. A total score is calculated by taking the average of responses and ranges from 0 to 4 where higher scores indicate greater use of strategies to lose or maintain weight.
Time Frame: Baseline and month 6
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From baseline to post-intervention (Month 6)
Description: No data was collected from the support group. Adverse event data was collected only on the participants.
Arm/Group | Participants
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT05275231/Prot_SAP_001.pdf
  • Informed Consent Form (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT05275231/ICF_000.pdf